CLINICAL TRIAL: NCT07383675
Title: EHR-Based Risk Factors With Prediction Models for Tinnitus Subtypes: A Multicenter Cross-sectional Study
Brief Title: A Multicenter Cross-sectional Study on Tinnitus Subtypes and Risk Factors
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Chongqing Renpin ENT. Hospital, China (Unknown); Nanjing Renpin ENT. Hospital, China (Unknown); Chengdu Renpin ENT. Hospital, China (Unknown)
Responsible Party: Principal Investigator, Hongsheng Tan, professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: TSM-2026
Record Dates: First submitted 2026-01-04; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — This is an observational study and no samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational group — This is a multicenter, cross-sectional observational study using existing electronic health record data collected during routine clinical care.We will use retrospectively extracted electronic health record data from multiple otolaryngology specialty hospitals to identify risk factors and develop predictive models for tinnitus subtypes at a single index time point.

SUMMARY:
Tinnitus affects an estimated 10-15% of the global population and can substantially impair quality of life, yet clinically actionable approaches for subtype identification and risk stratification remain limited. This multicenter, cross-sectional observational study will use de-identified electronic health record (EHR) data from three otolaryngology specialty hospitals in China to address these gaps. All extracted data will be de-identified with direct identifiers removed, and privacy safeguards will be implemented in accordance with institutional policies and applicable regulations to protect patient confidentiality.

DETAILED DESCRIPTION:
Using a prespecified, clinically informed framework, we will classify tinnitus into relevant subtypes, including somatosensory tinnitus, acute vs. chronic tinnitus, pulsatile tinnitus, and sudden hearing loss-related tinnitus. We will first describe the distribution of these subtypes and characterize their demographic, clinical, and laboratory profiles. We will then evaluate associations between candidate risk factors and subtype membership using multivariable analyses to quantify adjusted effects. Finally, we will develop and validate multivariable prediction models using both conventional statistical approaches and machine learning methods to support tinnitus subtype classification. Model performance will be assessed using discrimination, calibration, and clinical utility metrics. By integrating routine clinical data with biomarker information captured in real-world care, this study aims to provide evidence-based tools to improve tinnitus subtype diagnosis and enable more personalized clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old；
* Patients diagnosed with various types of tinnitus；
* Patients with available electronic medical records, including demographic and clinical information.

Exclusion Criteria:

* Patients with incomplete data；
* Patients with severe neurological；
* Patients with disorders that may confound tinnitus assessment.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any type of tinnitus from three otolaryngology specialty hospitals in China
Sampling Method: Non-Probability Sample
Enrollment: 3345 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Number of Patients in Each Tinnitus Subtype | baseline
  The number of participants classified into each predefined tinnitus subtype based on an integrated diagnosis clinical classification framework.

SECONDARY OUTCOMES:
Adjusted odds ratios of risk factors associated with each tinnitus subtype | baseline
  Multivariable logistic regression-derived odds ratios quantifying the independent association between risk factors and specific tinnitus subtypes.
Accuracy of prediction models for identifying tinnitus subtype classification | baseline
  The diagnostic performance of a multimodal classification model for identifying tinnitus subtype. The model integrates clinical characteristics, laboratory parameters, and computed tomography imaging features. Tinnitus subtype, determined by physician medical diagnosis, serves as the reference standard. Model performance will be quantified using the area under the receiver operating characteristic curve (AUC). The unit of measure is Area under the ROC curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Hongsheng Tan, Dr, Principal Investigator — Shanghai Jiao Tong University School of Medicne
Locations (1):
- Chongqing Renpin ENT Hospital, Chongqing, China